CLINICAL TRIAL: NCT01660061
Title: Monitoring Anticoagulant Therapy With Vitamin-K Antagonists in Patients With Antiphospholipid Syndrome
Brief Title: Monitoring Anticoagulant Therapy in Antiphospholipid Syndrome
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Birgit Linnemann, Priv.-Doz. Dr. Birgit Linnemann, Johann Wolfgang Goethe University Hospital
Other Study IDs: EV 77/11
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid syndrome; Antiphospholipid antibodies; Vitamin-K antagonists; International normalized ratio; Chromogenic factor X
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- APS patients: Patients with antiphospholipid syndrome requiring long-term anticoagulant therapy with vitamin-K antagonists
- Controls: Patients without antiphospholipid antibodies requiring anticoagulant therapy with vitamin-K antagonists

SUMMARY:
To Assess the Influence of Antiphospholipid Antibodies on INR Test Results in Patients with the Antiphospholipid Syndrome Anticoagulated with Vitamin-K Antagonists.

DETAILED DESCRIPTION:
Patients with an antiphospholipid syndrome receiving Vitamin-K antagonists for secondary prevention after a first thrombotic complication are known to be at higher risk of recurrent thrombotic events despite INR values in the therapeutic range. It ist also known that antiphospholipid antibodies can interfere with phospholipid-dependent tests (e.g. prothrombin time and INR).

The primary objective of this study is to determine the prevalence of interfering antiphospholipid antibodies. The intensity of anticoagulant therapy was assessed by measuring the INR using different thromboplastins and the CoaguChek system for INR self-assessment. Test results were compared to measurements of the phospholipid-independent chromogenic factor X.

The second objective of this study is to evaluate the incidence of recurrent thrombotic events during 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90 years

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with antiphospholipid syndrome requiring long-term treatment with vitamin-K antagonists (N=40) Pateints without antiphospholipid antibodies treated with vitamin-K antagonists (N=100)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference between INR and CFX correlate >20% | 0, 1, 2, 3, 6 and 12 month

SECONDARY OUTCOMES:
Arterial or venous thrombosis | 12 months
  Any arterial of venous thrombosis occurring under anticoagulant treatment with vitamin-K antagonists during 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Linnemann, MD, Principal Investigator — Goethe University Hospital, Division of Vascular Medicine
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- See also: Click here for more information about this study: Monitoring Anticoagulant Therapy in Antiphospholipid Syndrome — http://www.gefaesszentrum-frankfurt.de/forschung.php